CLINICAL TRIAL: NCT03967613
Title: Impact of an Intervention Based on a Multichannel Functional Electrical Stimulation (FES) Prototype on the Upper Limb Movement Quality in Post Stroke Patients
Brief Title: Functional Eletrical Stimulation in Post Stroke Patients
Acronym: FES-ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Allied Health Sciences of Porto (ESTSP) - Polytechnic Institute of Porto (IPP) (Other)
Collaborators: Fundación General CSIC (Unknown); Center for Rehabilitation Research (CIR) (Unknown); Tecnalia (Unknown)
Responsible Party: Principal Investigator, Rubim Santos, Rubim Santos, Polytechnic Institute of Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0348/CIE/ 6_E
Record Dates: First submitted 2018-12-18; First posted 2019-05-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: Functional eletrical stimulation; Stroke; Upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES (Experimental): Functional Eletrical Stimulation
  Interventions: Device: Functional eletrical stimulation

INTERVENTIONS:
Device: Functional eletrical stimulation — Aplication of functional eletrical stimulation on contralesional upper limb during functional tasks

SUMMARY:
The FES-ABLE project results from an Iberian partnership and aims to evaluate the impact of an intervention based on a functional electrical stimulation (FES) prototype on the upper limb movement quality during functional tasks. The results of this project will contribute to the definition of the therapeutic window of FES to improve upper limb function in stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* First and unilateral ischemic or hemorrhagic stroke, in the middle cerebral artery, confirmed by imaging;
* Age equal ou greater than 30 years old;
* Preserved congnitive function, corresponding to a score higher than 23 in the Mini Mental State Examination (MMSE);
* Ability to perform active movement in the contralesional upper limb (UL) of at least 15° in the shoulder and elbow.

Exclusion Criteria:

* Body mass index (BMI) less than 18,5 and greater than 30;
* Hemi-spatial neglect and/or uncorrected visual changes;
* Musculoskeletal or neurological conditions which may affect ULs and/or trunk function;
* Pain in the ULs;
* Severe sensorimotor impairment, corresponding to a score less than 39 in the Fugl-Meyer Assessment Scale - Upper Extremity (FMAS-UE);
* Lesions on the skin of the affected forearm;
* Severe spasticity (modified Ashworth >3);
* Severe muscle contractures on the affected forearm;
* Pacemaker;
* Osteosynthesis or metallic implants;
* Pregnancy;
* Adverse skin reaction to electrodes' gel.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Kinematic metrics change | Kinematic metrics will be assessed during 2 months and they will be reported through study completion, an average of 6 months
  End-point kinematics and joint kinematics will be analyzed. Regarding end-point kinematics, to evaluate speed, the absolute and relative movement times will be calculated separately for each phase and for the entire tasks, as well as the peak velocity for reach, forward and backward transport and return phases. To assess efficiency, smoothness and control strategy of movement, the índex of curvature, the number of velocity peaks (or number of motor units) and the time to peak velocity will be respectively calculated for reach, forward and backward transport and return phases.
  Regarding joint kinematics, joint angles5 of shoulder, elbow and wrist at onset of each phase will be calculated, as well as maximum aperture and time to maximum aperture in reach and return phases, and trunk displacement (to measure compensation) for each phase.

SECONDARY OUTCOMES:
User satisfaction | User satisfaction will be assessed during 2 months and it will be reported through study completion, an average of 6 months
  Participants' satisfaction will be assessed through an adaptation of the Reduced Upper Extremity Motor Activity Log Questionnaire. In this adapted questionnaire, the participant will be asked to classify the use of the arm in function of the quantity (0 - not used;1 - very rarely; 2 - rarely; 3 -half pre-stroke; 4- 3/4 pre-stroke; 5 - same as pre-stroke.) and quality (0 - not used.1 - very poor.2 - poor.3 - fair.4 - almost normal.5 - normal.) in the evaluated tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation Research, Porto, Portugal

REFERENCES:
- [Derived] Sousa ASP, Mesquita IA, Costa da Silva CI, Silva A, Macedo R, Imatz-Ojanguren E, Hernandez E, Keller T, Moreira J, Pereira da Fonseca PF, Santos R. Optimal Multifield Functional Electrical Stimulation Parameters for the "Turn on the Light" Task and Related Upper Limb Kinematics Repeatability in Poststroke Subjects. Arch Phys Med Rehabil. 2021 Jun;102(6):1180-1190. doi: 10.1016/j.apmr.2020.10.135. Epub 2020 Nov 27. PMID 33253692